CLINICAL TRIAL: NCT04261322
Title: Effect of X-ray on Rabies Virus in Vivo
Brief Title: Rabies Treatment by Exposure of Patient to X-Ray
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute For Research On Endemic Diseases And Liver, Egypt (Other Government)
Responsible Party: Principal Investigator, Ahmed Samir Mohammed El Behwashy, Principal Investigator, National Institute For Research On Endemic Diseases And Liver, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X-Ray as a treatment of Rabies
Record Dates: First submitted 2020-01-13; First posted 2020-02-07 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Treatment of Rabies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- rabies patient 1 (Experimental): not received immunoglobulins and symptomatic
  Interventions: Radiation: x ray exposure
- rabies patient 2 (Experimental): received immunoglobulins and symptomatic
  Interventions: Radiation: x ray exposure
- rabies patient 3 (Experimental): not received immunoglobulins and not yet symptomatic
  Interventions: Radiation: x ray exposure
- rabies patient 4 (Experimental): received immunoglobulins and not symptomatic
  Interventions: Radiation: x ray exposure

INTERVENTIONS:
Radiation: x ray exposure — exposure of whole body to x ray

SUMMARY:
x-ray has been proven to kill Rabies virus in vitro, so the investigators can use it in treatment of rabies infected patients.

DETAILED DESCRIPTION:
x-ray has been proven to kill Rabies virus in vitro, so the investigators can use it in treatment of rabies infected patients.

this can be done by exposure of infected , manifested patient who didn't receive prophylaxis or delayed in receiving immunoglobulins .

also can be applied to patients who have the injury in upper body near the CNS..

it's just an idea and the investigators need help to approve its effect and the investigators believe it will really work and give a new, rapid , cheap and very effective treatment to a 100% fatal disease..

the investigator also predict good results when x ray applied to some localized infections beside its current lines of treatment..

ELIGIBILITY:
Inclusion Criteria:

* patient bitten by rabid animal with signs and symptoms

Exclusion Criteria:

* bitten by non rabid animal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
the number of rabies infected, symptomatic patients who survived after x-ray exposure | 7 month
  detecting effect of x-ray exposure on treating Rabies

IPD SHARING:
Plan to Share IPD: Undecided